CLINICAL TRIAL: NCT02472184
Title: Office Based Evaluation of Patients Presenting With Abnormal Uterine Bleeding and/or Uterine Fibroids With Concurrent Office Hysteroscopy and Endometrial Biopsy; Does the Order Matter?
Brief Title: Optimal Order of Concurrent Office Hysteroscopy and Endometrial Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00022436
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2016-12

CONDITIONS: Uterine Fibroids; Vaginal Bleeding
Keywords: Office hysteroscopy; Endometrial biopsy; Abnormal uterine bleeding; Uterine fibroids
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage; Metrorrhagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Office Hysteroscopy (Active Comparator): Group of patients in which office hysteroscopy will be performed prior to endometrial biopsy
  Interventions: Procedure: Office hysteroscopy; Procedure: Endometrial biopsy
- Endometrial biopsy (Active Comparator): Group of patients in which endometrial biopsy will be performed prior to office hysteroscopy
  Interventions: Procedure: Office hysteroscopy; Procedure: Endometrial biopsy

INTERVENTIONS:
Procedure: Office hysteroscopy — Office hysteroscopy is a procedure performed in the office in which a flexible hysteroscope is inserted into the uterine cavity. The patient is positioned in a dorsal lithotomy position and teh cervix is visualized with a speculum. Normal saline is used to distend the cavity, and the hysteroscope is used to visualize any abnormalities within the cavity.
Procedure: Endometrial biopsy — An endometrial biopsy is a procedure in which a pipelle instrument is inserted into the uterine cavity and suction from the pipelle is used to obtain endometrial tissue. This is performed with the patient in the dorsal lithotomy position and a speculum is used to visualize the cervix.

SUMMARY:
This study will look at the optimal order in which to perform concurrent office hysteroscopy and endometrial biopsy in female patients who present for evaluation of abnormal uterine bleeding at a fibroid and endometriosis treatment center.

DETAILED DESCRIPTION:
This will be a prospective single blinded randomized control trial to determine whether the order of performance of office hysteroscopy (OH) and endometrial biopsy (EMB) during the same office evaluation for abnormal uterine bleeding affects the patient's pain perception. We also intend to investigate whether the order of the procedures affects the adequacy of the endometrial sample, duration of the procedure, and optimal visualization of the uterine cavity. We hypothesize that performing EMB prior to OH will result in higher patient pain scores.

Included patients will be all consecutive female patients ages 18-70 presenting to the University of South Florida Center for Endometriosis and Fibroid Treatment (CFERT) for evaluation of abnormal uterine bleeding or uterine fibroids.

Patients will be randomly assigned to have either OH followed by EMB or EMB followed by OH as part of their clinical assessment of AUB/uterine fibroid based on clinical indication. The patients will be informed about the two indicated procedures by their clinical provider but will be blinded to the order of performance. The healthcare provider/investigator will be aware of the order in which the procedures are assigned and to be performed. Patients will be consented to participate in the study prior to the procedure by the study team on the day the indicated procedures are scheduled in CFERT. The healthcare provider performing the procedure will open an unlabeled envelope, within which there will be a piece of paper indicating which procedure is to be performed first. This will then be recorded in the study log. The study log will include enrolled patients, assigned study number which will range from 001 to the minimum number of patients required for the study as indicated by sample size calculation.

At the end of the procedures, patient will be asked to describe their pain perception based on Visual analogue scale (VAS) from 0-10. The adequacy of the endometrial sample will be determined from the pathology report. The duration of the entire procedures (min) will be timed using a stopwatch from the time of insertion of the hysteroscope/Pipelle catheter in the external cervical canal to removal of the instruments. A panoramic picture of the endometrial cavity will be taken and will be given to a blinded independent reviewer to determine the adequacy of visualization based on 3 point scoring system (fair, good and excellent). Fair visualization will be defined as no tubal ostia visualized; good will be defined as both tubal ostia identified but only able to visualize 180 degrees of panorama; excellent visualization will be defined as visualizing bilateral tubal ostia and having a clear image of the uterine cavity in 360 degrees of panorama.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive female patients ages 18-70 presenting to the Center for Fibroid and Endometriosis Research and Treatment for medically indicated office hysteroscopy and endometrial biopsy for evaluation of abnormal uterine bleeding and or uterine fibroids with ability to provide written informed consent.

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients presenting to the Center for Fibroid and Endometriosis Research and Treatment for medically indicated office hysteroscopy and endometrial biopsy for evaluation of abnormal uterine bleeding and or uterine fibroids are not deemed clinically indicated based on the assessment of their clinical provider.
* Patients in which office hysteroscopy or endometrial biopsy is unsuccessful due to patient discomfort, known cervical stenosis, or poor visualization of the cervix

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Patient pain scores | Immediately following procedures
  After the procedures are performed, the patient will be asked to describe their pain perception based on Visual analogue scale (VAS) from 0-10

SECONDARY OUTCOMES:
Adequacy of endometrial sample | Within 2 weeks following endometrial biopsy
  The adequacy of the endometrial sample will be determined from the pathology report.
Duration of procedure | Immediately following procedure
  The duration of the entire procedures (min) will be timed using a stopwatch from the time of insertion of the hysteroscope/Pipelle catheter in the external cervical canal to removal of the instruments.
Visualization of endometrial cavity | During procedure
  A panoramic picture of the endometrial cavity will be taken and will be given to a blinded independent reviewer to determine the adequacy of visualization based on 3 point scoring system (fair, good and excellent). Fair visualization will be defined as no tubal ostia visualized; good will be defined as both tubal ostia identified but only able to visualize 180 degrees of panorama; excellent visualization will be defined as visualizing bilateral tubal ostia and having a clear image of the uterine cavity in 360 degrees of panorama.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Imudia, MD, Principal Investigator — University of South Florida College of Medicine Department of Infertility and Reproductive Endocrinology
Locations (1):
- University of South Florida College of Medicien Department of Obstetrics and Gynecology, Tampa, Florida, United States

REFERENCES:
- [Background] Committee on Practice Bulletins-Gynecology. Practice bulletin no. 128: diagnosis of abnormal uterine bleeding in reproductive-aged women. Obstet Gynecol. 2012 Jul;120(1):197-206. doi: 10.1097/AOG.0b013e318262e320. No abstract available. PMID 22914421
- [Background] Technology assessment No. 7: Hysteroscopy. Obstet Gynecol. 2011 Jun;117(6):1486-1491. doi: 10.1097/AOG.0b013e3182238c7d. PMID 21606772
- [Background] Kelekci S, Kaya E, Alan M, Alan Y, Bilge U, Mollamahmutoglu L. Comparison of transvaginal sonography, saline infusion sonography, and office hysteroscopy in reproductive-aged women with or without abnormal uterine bleeding. Fertil Steril. 2005 Sep;84(3):682-6. doi: 10.1016/j.fertnstert.2005.03.036. PMID 16169403
- [Background] Clark TJ, Voit D, Gupta JK, Hyde C, Song F, Khan KS. Accuracy of hysteroscopy in the diagnosis of endometrial cancer and hyperplasia: a systematic quantitative review. JAMA. 2002 Oct 2;288(13):1610-21. doi: 10.1001/jama.288.13.1610. PMID 12350192
- [Background] Ghaly S, de Abreu Lourenco R, Abbott JA. Audit of endometrial biopsy at outpatient hysteroscopy. Aust N Z J Obstet Gynaecol. 2008 Apr;48(2):202-6. doi: 10.1111/j.1479-828X.2008.00834.x. PMID 18366496
- [Derived] Sarkar P, Mikhail E, Schickler R, Plosker S, Imudia AN. Optimal Order of Successive Office Hysteroscopy and Endometrial Biopsy for the Evaluation of Abnormal Uterine Bleeding: A Randomized Controlled Trial. Obstet Gynecol. 2017 Sep;130(3):565-572. doi: 10.1097/AOG.0000000000002202. PMID 28796688